CLINICAL TRIAL: NCT06505291
Title: Long-term Management of Patients With Ruptured HCC
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: CHCrompu
Record Dates: First submitted 2024-06-25; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 16 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this work is to evaluate the prevalence and results of specific management of HCC after spontaneous rupture, since the arrival of sorafenib in 2008.

DETAILED DESCRIPTION:
Retrospective, observational, multicenter study over the period from January 2008 to April 2024.

Cases had to be 18 years or older. They were identified by two different methodologies adapted to the 4 participating centers. In particular, a request for ICD10 C22.0 (CHC) codes associated with K66.1 (hemoperitoneum) was carried out by the medical information departments (DIM) of the Caen University Hospital and the Avicenne hospital. Secondly, the automated keyword selection tools "Cohort 360" and "i2b2" were used at the La Pitié Salpetrière and Paul Brousse hospital centers to identify the terms "CHC" and "ruptured" in the computerized patient files. Secondarily, duplicates and coding errors were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Ruptured hepatocellular carcinoma with or without cirrhosis

Exclusion Criteria:

* Liver adenoma without histologically proven HCC
* Other benign or malignant liver tumors
* ATCD of potentially triggering interventional procedure in the previous month.
* Hemorrhagic ascites without tumor
* Intratumoral hemorrhages without hemoperitoneum or capsular rupture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with ruptured hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Survival after rupture of hepatocellular carcinoma | 15 years

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Commin A, Metivier C, Allaire M, Lubrano J, Claudinot A, Coilly A, Allard MA, Roux C, Scatton O, Nault JC, Sutter O, Ganne-Carrie N, Ngo TV, Goff VL, Ali ZB, Tedlaouti H, Papin J, Habireche M, Lebedel L, Perignon C, Dao T, Morello R, Ollivier-Hourmand I. Early Hemostatic Treatment Could Improve 30-Day Survival After Spontaneous Rupture of Hepatocellular Carcinoma. Liver Int. 2025 Oct;45(10):e70332. doi: 10.1111/liv.70332. PMID 40990229